CLINICAL TRIAL: NCT04124861
Title: Evaluation and Prediction of Relapse Risk After Glucocorticoid and Immunosuppressant Withdrawal in Patients With Stable IgG4 Related Disease: An Open-labeled Multi-centric Randomized Controlled Study From China
Brief Title: Withdraw Drug in Stable IgG4-Related Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Peking University People's Hospital (Other); The People's Hospital of Hebei Province (Other); Shengjing Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Withdraw drug in IgG4-RD
Record Dates: First submitted 2019-02-13; First posted 2019-10-11 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Autoimmune Diseases
Keywords: Immunoglobulin G4-Related Disease
MeSH Terms: conditions — Autoimmune Diseases; Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug free (Experimental): Arm A: Drug free Glucocorticoid（GC）is tapered and stopped in 8 weeks(GCs at a dose of ≤ 2.5 mg of prednisone or equivalent for treatment of adrenal insufficiency) .
  Immunosuppressant is also tapered and discontinues in 8 weeks.
  Interventions: Drug: Drug free, IS monotherapy and GC combined with IS
- IS monotherapy (Experimental): Arm B: Immunosuppressant only Glucocorticoid（GC）is tapered and stopped in 8 weeks. The same type and dosage of immunosuppressive agent before admission, including Mycophenolate mate(<= 1g/d) or Leflunomide (<=20mg/d) or Methotrexate (<=15mg/w) or Azathioprine (<=100mg/d)
  Interventions: Drug: Drug free, IS monotherapy and GC combined with IS
- GC combined with IS (Experimental): Arm C: GC+Immunosuppressant Both Glucocorticoid(GC) (no more than 7.5mg/d) and immunosuppressant are kept as maintaining dose.
  Interventions: Drug: Drug free, IS monotherapy and GC combined with IS

INTERVENTIONS:
Drug: Drug free, IS monotherapy and GC combined with IS — Follow-up intervals: Every 3 months (3th, 6th, 9th, 12th, 15th, 18th month).

SUMMARY:
Evaluation and prediction of relapse risk after glucocorticoid or immunosuppressant withdrawal in patients with stable IgG4 related disease: a prospective cohort study from china.

DETAILED DESCRIPTION:
IgG4-related disease (IgG4-RD) is a chronic autoimmune disease with a relapsing-remitting course. For patients in remission, glucocorticoid (GC) and immunosuppressant are used to be maintained for a long time in fear of disease flare. Long-term GC and immunosuppressant could bring a lot of side-effects and economic burden. Whether and when patients with stable disease should withdraw GC or immunosuppressant? How about the relapse risk respectively? What are the risk factors for disease flare? All the above remain unclear. The aim of this study is to explore the relapse risk after GC or immunosuppressant withdrawal in IgG4-RD patients with stable disease and to establish a predictive model for risk stratification. Meanwhile the investigators aim to testify the effects of immunosuppressant in preventing IgG4-RD relapse. This study is a prospective cohort clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must meet the following diagnostic criteria of IgG4RD (2011): 1)Swelling, sclerosing and inflammatory involvement of one or more organ, including sclerosing pancreatitis, sialadenitis (Mikulicz disease), sclerosing cholangitis, inflammatory pseudotumors, retroperitoneal or mediastinal fibrosis, interstitial nephritis, hypophysitis, sclerosing dacryoadenitis, inflammatory aortic aneurysm, lymphadenopathy, or other inflammatory conditions; 2)Elevated serum IgG4 (>1.35 g/L); 3)Histopathologic features of fibrosis and/or lymphocytic and polyclonal plasma cell infiltration (and IgG4+ plasma cells on immunohistology when performed). Patients fulfill 1)+2)+3) are diagnosed as definite IgD4RD, 1)+2): possible IgG4RD; 1)+3): probable IgG4RD. exclusion of other diseases.
2. Disease stabilized more than one year (Responder Index < 2 points)
3. Dose of Glucocorticoid(GC): prednisone (or equivalent) ≤ 7.5mg/d for more than 6 months
4. Immunosuppressant: one of the following drugs, the same dose maintain at least 3 months (Mycophenolate mate <= 1g/d or Leflunomide <=20mg/d or Methotrexate <=12.5mg/w or Azathioprine <=100mg/d).

Exclusion Criteria:

1. Patient was diagnosed other connective tissue diseases
2. Patient with tumor
3. Women during pregnancy or planning pregnancy
4. Patient with active infections, including HIV, HCV, HBV, TB, etc.
5. Patient with severe irreversible organ damage
6. Active IgG4-RD, responder index >= 2 points
7. Stable condition less than one year.
8. Patient with two or more immunosuppressive agents.
9. Biological agents (such as CD20 monoclonal antibody and TNF-a inhibitor) have been used for half a year before admission.
10. Patient with IgG4-RD recurrence during hormone reduction in the past.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The difference of recurrent rate of IgG4-RD among three groups. | One and half year
  Clinical recurrence definition: any item of IgG4-RD Responder Index >=2，new organ involvement; with or without elevated serum IgG4 levels. Serum recurrence definition: Serum IgG4 level was higher than baseline level, IgG4-RD Responder Index was higher than or equal to 1 point, without clinical symptom or imaging deterioration.

SECONDARY OUTCOMES:
The changes of IgG4-RD Responder Index | One and half year
  According to IgG4-RD responder Index Validation Study (Version: 13, December, 2015)
The changes of serum IgG4 levels | One and half year
  Level of serum IgG4(mg/dL)
The changes of serum IgG level | One and half year
  Level of serum IgG(g/L)
The changes of serum hsCRP level | One and half year
  Level of serum high-sensitivity C-reactive protein level(mg/L)
The changes of ESR | One and half year
  Serum erythrocyte sedimentation rate(mm/h)
The percentages of adverse events | One and half year
  Adverse effect of drugs

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD., Principal Investigator — Peking Union Medical College Hospital; Yunyun Fei, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Peng L, Nie Y, Zhou J, Wu L, Chen X, Wang F, Li J, Peng Y, Lu H, Zhao L, Li M, Zhao Y, Zeng X, Fei Y, Zhang W. Withdrawal of immunosuppressants and low-dose steroids in patients with stable IgG4-RD (WInS IgG4-RD): an investigator-initiated, multicentre, open-label, randomised controlled trial. Ann Rheum Dis. 2024 Apr 11;83(5):651-660. doi: 10.1136/ard-2023-224487. PMID 38216319